CLINICAL TRIAL: NCT04888858
Title: Effect of Epidural Analgesia During Labor on Force of Maternal Push
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The PI, Dr. Younger, left Henry Ford Health.
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Katherine Nowak, Senior Staff Anesthesiologist, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 14173
Record Dates: First submitted 2021-05-06; First posted 2021-05-17 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Labor Pain; Analgesia; Maternal; Procedure
MeSH Terms: conditions — Labor Pain; Agnosia | interventions — Analgesia, Epidural

STUDY DESIGN:
Intervention Model Description: The force of the maternal push when performing Valsalva maneuver will be compared before and after administration of epidural analgesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Epidural Analgesia (Experimental): All subjects will be given epidural analgesia to treat their labor pain. As part of standard protocol for all patients who receive a labor epidural, the epidural will then be tested using 3ml of 1.5% lidocaine and 1:200,000 epinephrine test solution, and the epidural catheter will then be loaded with 10ml of 0.125% bupivacaine solution. The epidural catheter will then be connected to a programmed intermittent epidural bolus pump which will administer 5ml of a 0.125% bupivacaine/2mcg fentanyl solution every 30minutes. The first dose will be given following 30minutes after the loading dose. 30 minutes after loading the loading dose and after the first pump dose has been given, we will assess the VAS pain scores and the level of the analgesic based on decreased sensation to ice.
  Interventions: Drug: Epidural analgesia (0.125% bupivacaine/2mcg fentanyl solution)

INTERVENTIONS:
Drug: Epidural analgesia (0.125% bupivacaine/2mcg fentanyl solution) — As part of standard protocol for all patients who receive a labor epidural, the epidural will then be tested using 3ml of 1.5% lidocaine and 1:200,000 epinephrine test solution, and the epidural catheter will then be loaded with 10ml of 0.125% bupivacaine solution. The epidural catheter will then be connected to a programmed intermittent epidural bolus pump which will administer 5ml of a 0.125% bupivacaine/2mcg fentanyl solution every 30minutes. The first dose will be given following 30minutes after the loading dose. 30 minutes after loading the loading dose and after the first pump dose has been given, we will assess the VAS pain scores and the level of the analgesic based on decreased sensation to ice.

SUMMARY:
There are multiple factors that determine progress of normal vaginal delivery. Frequency, duration and strength of uterine contractions are important for progress throughout labor, and abdominal wall muscle contractions contribute to progress during the final stage. Epidural analgesia helps to alleviate the pain associated with uterine contractions, this however this comes at the expense of prolonging labor by reducing the strength of abdominal wall muscle contractions.

The purpose of this prospective study is to quantify how much epidurals decrease the strength of abdominal wall contractions. Intraabdominal pressure will be used as surrogate to strength of abdominal wall contractions, and it will be measured via a foley catheter inserted into the urinary bladder as part of standard procedure for patients receiving labor epidurals. We will compare the change in intraabdominal pressure when patients perform forceful abdominal contractions (valsalva maneuvers) prior to and during epidural analgesia. This will lay the foundation for a future study in which we plan to compare the effects of different epidural analgesia types and concentrations on abdominal wall muscle contractions.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years and older)
* Pregnant women in their third trimester
* Able to read and speak English
* Capacity to consent to participate
* Receiving a labor epidural catheter during their labor and delivery at HFH-Main

Exclusion Criteria:

* Severe cardiac disease
* People who are unable/medically recommended not to perform valsalva maneuvers
* People who are not undergoing labor epidural analgesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients must be healthy pregnant women that have reached the decision to receive epidural analgesia for their labor.
Enrollment: 0 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-07-02 (Actual); Study Completion 2022-07-02 (Actual)

PRIMARY OUTCOMES:
The change in intraabdominal pressure (surrogate of maternal force) | 2 hours following initial administration of labor epidural
  The change in intraabdominal pressure will be measured prior to receiving epidural analgesia, and again at 1 and 2 hours following administration. The change observed before and after will be compared to quantify the decreased change following epidural administration.

SECONDARY OUTCOMES:
Mode of delivery | Up to 72 hours after initial administration of labor epidural
  Whether the child is delivered via vaginal or cesarean birth.
Duration of second stage of labor | Up to 72 hours after initial administration of labor epidural
  How long the second stage of labor takes.
Apgar scores | Up to 72 hours after initial administration of labor epidural
  The apgar scores will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to share individual participant data with other researchers.